CLINICAL TRIAL: NCT02263417
Title: The Safety and Efficacy of Long-term Treatment of PINS Stimulator System for Patients With Dystonia
Brief Title: A Randomized Controlled Trail Comparing Subthalamic and Pallidal Deep Brain Stimulation for Dystonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Pins Medical Co., Ltd (Industry)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PINS-005
Record Dates: First submitted 2014-09-27; First posted 2014-10-13 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Dystonia
MeSH Terms: conditions — Dystonia | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep Brain Stimulation (Active Comparator): Stimulation is on
  Interventions: Device: Deep Brain Stimulation (DBS) of Gpi; Device: Deep Brain Stimulation (DBS) of STN
- Placebo (Sham Comparator): Stimulation is off
  Interventions: Device: Deep Brain Stimulation (DBS) of Gpi; Device: Deep Brain Stimulation (DBS) of STN

INTERVENTIONS:
Device: Deep Brain Stimulation (DBS) of Gpi
  Other Names: Rechargeable Neurostimulator
Device: Deep Brain Stimulation (DBS) of STN
  Other Names: Rechargeable Neurostimulator

SUMMARY:
The purpose of this study was to compare the subthalamic nucleus(STN) with the globus pallidus internus(GPi) as a stimulation target for deep brian stimulation(DBS) for medically refractory dystonia.

DETAILED DESCRIPTION:
In this prospective randomized controlled study,elecrodes were bilaterally implanted in STN and Gpi of 40 patients with dystonia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18 to 75 years old, male or female.
2. Diagnosed with cervical dystonia by a movement disorders neurologist.
3. Has cervical dystonia alone, not generalized or multifocal.
4. Has had adequate trials of medical therapy.

Exclusion Criteria:

1. Cognitive impairment.
2. Abnormalities on pre-operative magnetic resonance imaging (MRI).
3. Medical conditions precluding general anaesthetic or surgery.
4. Unstable psychiatric disease.
5. Previous brain lesions to treat cervical dystonia.
6. Attended some other trials within three month.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-07; Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Burke-Fahn-Marsden Scale (BFM) | Change from baseline in BMF at 1, 3 months and 6 months

SECONDARY OUTCOMES:
Quality of life (SF-36) | Change from baseline in SF-36 at 1, 3 months and 6 months
Psychiatric assessment (HADS-D and PANSS) | Change from baseline in HADS-D and PANSS at 1, 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Luming, PhD, Study Chair — Tsinghua University
Locations (1):
- Peking union medical college hospital, Beijing, Beijing Municipality, China